CLINICAL TRIAL: NCT02496520
Title: Dendritic Cell-based Immunotherapy for Advanced Solid Tumours of Children and Young Adults
Acronym: DEND/TIA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEND/TIA; 2013-003632-71 (EudraCT Number)
Record Dates: First submitted 2015-06-15; First posted 2015-07-14 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2019-05

CONDITIONS: Sarcoma; Central Nervous System Tumor
Keywords: dendritic cell vaccination; sarcoma; central nervous system tumor; childhood; adolescent; immunotherapy
MeSH Terms: conditions — Sarcoma; Central Nervous System Neoplasms | interventions — Surgical Procedures, Operative; Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccines with autologous dendritic cells (Experimental): Vaccines with autologous dendritic cells
  Interventions: Biological: dendritic cells; Procedure: Surgery as needed by the patient´s tumor and stage; Drug: Chemotherapy as needed by the patient´s tumor and stage; Radiation: Radiation therapy as needed by the patient´s tumor and stage

INTERVENTIONS:
Biological: dendritic cells — vaccines with dendritic cells pulsed with tumor lysate
Procedure: Surgery as needed by the patient´s tumor and stage
Drug: Chemotherapy as needed by the patient´s tumor and stage
Radiation: Radiation therapy as needed by the patient´s tumor and stage

SUMMARY:
Phase I/II, open, prospective clinical trial, historically controlled. The objective is to evaluate the safety and, as a secondary measure, the efficacy of an experimental treatment based on a cellular therapy (vaccination with autologous dendritic cells pulsed with tumor lysate) in patients affected of metastatic or relapsed sarcomas or (Central Nervous System) CNS tumors.

DETAILED DESCRIPTION:
Phase I/II, open, prospective clinical trial, historically controlled. Patients affected of metastatic or relapsed sarcomas or (Central Nervous System) CNS tumors will be included. The patients will receive standard treatment and experimental treatment based on a cellular therapy with vaccination with autologous dendritic cells pulsed with tumor lysate. The immunization schedule includes 4 monthly vaccines, 4 bimonthly and quarterly remaining vaccines. The vaccines will be administered intradermally in combination with standard treatment for each type of tumor.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosis or metastatic or relapsed sarcoma or high grade central nervous system tumor
* From 3 to 40 years
* Surgery feasibility. In the central nervous system tumors, residual tumor after surgery must be minimal.

Exclusion Criteria:

* Toxicity or liver, medullar, renal insufficiency that advise against participation
* Pregnant or breast feeding women
* Diagnosis of other tumor than basal cell squamous carcinoma of the skin or in situ cervix carcinoma
* Immunosuppressive treatment
* Human Immunodeficiency virus (HIV), hepatitis B, hepatitis C or syphilis infection

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2018-09-16 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Number and type of adverse events detected in the follow up as a measure of safety and tolerability | 24 months

SECONDARY OUTCOMES:
Event free progression, overall survival, time to progression and number and size of existent tumoral lesions as measures of clinical efficacy | 36 months
Humoral and cellular immune response as a measure of the immunogenicity of the vaccine. | 2 weeks to 24 months
Quality of life measured with QLQ-C30, QLQ-BN20 questionnaires. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Ana Patiño-García, PhD, Principal Investigator — CUN
Locations (1):
- University Clinic of Navarra, Pamplona, Navarre, Spain